CLINICAL TRIAL: NCT00709267
Title: A Randomized, Open Label Absolute Bioavailability Study of Folic Acid.
Brief Title: Bioavailability Study of Folic Acid in Healthy Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CR002386
Record Dates: First submitted 2008-06-30; First posted 2008-07-03 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Healthy; Pharmacokinetics
Keywords: Folic Acid; Chemistry, Analytical; Administration, Oral; Infusions, Intravenous; Biological Availability; Safety
MeSH Terms: interventions — Folic Acid

INTERVENTIONS:
Drug: Folic acid

SUMMARY:
The purpose of the study is to determine the bioavailability of orally administered folic acid compared with the i.v. administered folic acid, and to use the samples collected to validate the analytical methods for estimation of folic acid in plasma and red blood cells (RBCs).

DETAILED DESCRIPTION:
Few formal pharmacokinetic studies have been conducted with folic acid to determine its absolute bioavailability, pharmacokinetic profile, or intra- and intersubject variability. Moreover, most analytical work has been completed in academic settings, and no Good Laboratory Practice (GLP)-validated assay method has been developed. This was a randomized (study drug assigned by chance), open-label, 3-way crossover, single-center trial, consisting of a prerandomization phase, an open-label treatment phase (3 single doses separated by washouts of 7 days each), and a posttreatment phase. Healthy volunteers were randomly assigned to 1 of 6 treatment sequences (2 healthy volunteers per sequence). All healthy volunteers received a single dose of folic acid in each treatment period (400-mcg oral solution, 400-mcg i.v. infusion, and a 1-mg oral tablet). Blood samples for pharmacokinetic analysis were collected at specified times following each dose. Blood samples for measurement of red cell folate were collected before dosing on Day 1 of Period 1. For each period, healthy volunteers were confined to the study unit from the evening before Day 1 through the completion of the Day 2 assessments (24-hour pharmacokinetic blood sample collection). End-of-study assessments took place on Day 17 or at the time of early withdrawal. Safety was evaluated based on the monitoring of adverse events, vital sign measurements, physical examinations, and clinical laboratory tests. Heart rate and blood pressure were measured at screening, on the first day of each treatment period (Days 1, 8, and 15), and at study completion (Day 17) or early withdrawal; body temperature was measured at screening only. A physical examination was performed at screening and at study completion (Day 17) or early withdrawal. Blood samples for serum chemistry and hematology and a random urine sample for urinalysis were taken at the start of the study, Days -21 to -2, and at the end of the study (Day 17 or early termination).

All subjects received a single dose of folic acid in each treatment period (400-mcg oral solution, 400-mcg i.v. infusion, and a 1-mg oral tablet), separated by washouts of 7 days each.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Nonpregnant
* Nonlactating
* Nonsmoking women
* With a history of regular menstrual cycles
* Weighing at least 110 pounds
* Having a body mass index between 18 and 28 kg/m2
* And having a hematocrit of at least 36%

Exclusion Criteria:

* Known history of vitamin B-12 deficiency or a current need for vitamin B-12 injections
* Elevated blood pressure (BP) (i.e., sitting systolic BP >140 mm mercury [Hg] and/or diastolic BP >90 mm Hg)
* Had tested positive for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (anti-HCV)
* Recent history (within 12 months prior to the first admission visit) of alcohol or other substance abuse or tested positive for drugs of abuse, such as amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, and tricyclic antidepressant agents
* Used barbiturates, antiepileptics, rifampin, griseofulvin, St. John's Wort or other hepatic enzyme inducing drugs within 30 days before randomization

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2004-10; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Determine the absolute bioavailability of orally administered folic acid; Estimate intrasubject variance; Validate analytical methods to determine the folate levels in plasma and RBCs

SECONDARY OUTCOMES:
Assessment of safety

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Bioavailability study of folic acid in healthy women — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=476&filename=CR002386_CSR.pdf